CLINICAL TRIAL: NCT00992446
Title: Bortezomib* and Vorinostat as Maintenance Therapy After Autologous Transplant for Non-Hodgkin Lymphoma Using R-BEAM or BEAM Conditioning Transplant Regimen
Brief Title: Bortezomib and Vorinostat as Maintenance Therapy After Autologous Stem Cell Transplant in Treating Patients With Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leona Holmberg, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2292.00; NCI-2009-01302 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FH 2292/X05287 (Other: Fred Hutchinson Cancer Research Center); X05287; 2292.00 (Other: Fred Hutchinson Cancer Research Center); P30CA015704 (NIH)
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-02

CONDITIONS: Adult Diffuse Large B-Cell Lymphoma; B-Cell Non-Hodgkin Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Non-Hodgkin Lymphoma; T-Cell Non-Hodgkin Lymphoma
Keywords: Autologous stem cell transplant; NHL; maintenance therapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell | interventions — Bortezomib; Carmustine; carmustine, poliferprosan 20 drug combination; Cytarabine; Etoposide; Melphalan; Rituximab; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy, ASCT, bortezomib, vorinostat)) (Experimental): All patients receive carmustine IV over 3 hours on day -7; cytarabine IV BID over 3 hours and etoposide IV BID over 2 hours on days -6 to -3; and melphalan IV over 30 minutes on day -2. Only patients with history of CD20+ NHL receive additional rituximab IV on days -19 and -12. Patients undergo ASCT on day 0. Patients then receive bortezomib IV on days 2 and 8, and vorinostat PO QD on days 1-14. Treatment with bortezomib and vorinostat repeats for total of 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Bortezomib; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Drug: Melphalan; Drug: Rituximab; Drug: Vorinostat

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: Autologous Stem Cell Transplantation
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Rituximab — Given IV
  Other Names: BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar BI 695500; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; RTXM83
Drug: Vorinostat — Given PO
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial studies the side effects and how well bortezomib and vorinostat work in treating patients with non-Hodgkin lymphoma (NHL) after patients' own stem cell (autologous) transplant. Bortezomib and vorinostat in the laboratory may stop the growth of lymphoma cells and make them more likely to die by blocking some of the enzymes needed for cell growth. Giving bortezomib together with vorinostat after an autologous stem cell transplant may thus kill lymphoma cells that remain after transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess toxicities of combining vorinostat and bortezomib as maintenance therapy after autologous stem cell transplant (ASCT) for NHL.

SECONDARY OBJECTIVES:

I. Ability to complete planned therapy.

II. Time to disease progression, event-free survival.

III. Overall survival.

OUTLINE:

All patients receive carmustine intravenously (IV) over 3 hours on day -7; cytarabine IV twice daily (BID) over 3 hours and etoposide IV BID over 2 hours on days -6 to -3; and melphalan IV over 30 minutes on day -2. Only patients with history of cluster of differentiation (CD)20+ NHL receive additional rituximab IV on days -19 and -12. Patients undergo ASCT on day 0. Patients then receive bortezomib IV on days 2 and 8, and vorinostat orally (PO) once daily (QD) on days 1-14. Treatment with bortezomib and vorinostat repeats for total of 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA FOR AUTOLOGOUS TRANSPLANT
* Diagnosis of non-Hodgkin's lymphoma, transformed B-cell lymphoma, follicular lymphoma, mantle cell lymphoma, diffuse large B-cell or T-cell lymphoma, and deemed a candidate for autologous transplant
* American Heart Association class I: patients with cardiac disease but without resulting limitation of physical activity; ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain; additionally, patients > 60 years of age must have a left ventricular ejection fraction of at least >= 40% demonstrated by multi gated acquisition scan (MUGA) or echocardiogram (Echo)
* Total bilirubin =< 1.5 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x the upper limit of normal
* Creatinine clearance (CrCL) (calculated creatinine clearance is permitted) > 40 mL/min
* Diffusing capacity of the lung for carbon monoxide (DLCO), forced expiratory volume in one second (FEV1), and forced vital capacity (FVC) >= 50% of predicted (corrected for hemoglobin)
* Autologous graft with a minimum of >= 3.0 x 10^6 CD34+ cells/kg; not CD34 selected
* Signed informed consent
* Female patients of childbearing potential has a negative serum pregnancy test beta-human chorionic gonadotropin (hCG)
* Female patient is either postmenopausal, free from menses for >= 2 years, surgically sterilized, or willing to use 2 adequate barrier methods of contraception to prevent pregnancy or agrees to abstain from heterosexual activity throughout the study
* Male patient agrees to use an adequate method of contraception for the duration of the study
* INCLUSION CRITERIA FOR MAINTENANCE THERAPY
* 30-120 days post ASCT for non-Hodgkin's lymphoma
* CrCL >= 40 ml/min
* Platelets (PLT) >= 75,000 cells/mm^3 for 5 days after recovery from ASCT nadir
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 for 5 days after recovery from ASCT nadir
* Total bilirubin (TB) =< 1.5 x upper limit of normal (ULN)
* AST/ALT =< 2.5 x ULN

Exclusion Criteria:

* EXCLUSION CRITERIA FOR AUTOLOGOUS TRANSPLANT
* Karnofsky performance score < 70%
* Uncontrolled bacterial, viral, or fungal infection (currently taking medication and with progression or no clinical improvement)
* Pregnant or breastfeeding
* Fertile men and women unwilling to use contraceptive techniques from the time of transplant until one month post maintenance therapy
* Prior autologous or allogeneic hematopoietic stem cell transplantation (HSCT)
* Patients with evidence of myelodysplastic syndromes (MDS)/acute myeloid leukemia (AML) or abnormal cytogenetics analysis indicative of MDS on the pre-transplant bone marrow examination
* Prolonged corrected QT interval (QTC) on electrocardiogram (EKG)
* Poorly-controlled diabetes mellitus (DM)
* >= grade 2 peripheral neuropathy
* Prior history of human immunodeficiency virus (HIV) positivity or known history of hepatitis B or C
* Previous history of hypersensitivity to bortezomib, boron, or mannitol; known hypersensitivity to the components of study drug or its analogs
* Require therapeutic anticoagulation treatment, especially with Coumadin
* Patient who has had chemotherapy, radiotherapy, or biological therapy, within 30 days (42 days for nitrosoureas or mitomycin C) or who has not recovered from adverse events due to agents administered more than 30 days earlier
* Patient is currently participating or has participated in a study with an investigational compound or devise within 30 days of initial dosing with study drug(s)
* Patient had prior treatment with an histone deacetylase (HDAC) inhibitor (e.g., romidepsin [Depsipeptide], NSC-630176, MS 275, LAQ-824, belinostat [PXD-101], LBH589, MGCD0103, CRA024781, etc); patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study; patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period
* History of central nervous system (CNS) disease
* Symptomatic ascites or pleural effusions
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs, substance abuse or had a recent history (within the last year) of drug or alcohol abuse
* Patient with a history of a prior malignancy with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma or an in situ malignancy; adequately treated localized prostate carcinoma with prostate-specific antigen (PSA) < 1.0; or who has undergone potentially curative therapy with no evidence of disease for five years, and/or who is deemed at low risk for recurrence by his/her treating physician
* Patient has a history or current evidence of any condition, therapy, or laboratory (lab) abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient to participate
* Patient has a history of a gastrointestinal surgery or other procedures that might, in the opinion of the investigator, interfere with the absorption or swallowing of the study drugs
* EXCLUSION CRITERIA FOR MAINTENANCE THERAPY
* >= grade 2 peripheral neuropathy within 14 days before beginning maintenance therapy
* Prolonged QTC
* Poorly-controlled DM
* Myocardial infarction (MI) with ASCT or developed dilated cardiomyopathy with ASCT
* Untreated systemic infection
* Potassium (K) and magnesium (Mg) >= grade 2 toxicity
* Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Patient has hypersensitivity to VELCADE (bortezomib), boron, or mannitol
* Female subject is pregnant or lactating; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for postmenopausal or surgically sterilized women
* Female patients who are lactating or have a positive serum pregnancy test during the screening period, or a positive urine pregnancy test on day 1 before first dose of study drug, if applicable
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial
* Radiation therapy within 3 weeks before randomization; enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-09-02 (Actual); Primary Completion 2015-06-17 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat))
Started | 27
Completed | 19
Not Completed | 8
Not completed — Disease Progression | 1
Not completed — Withdrawal by Subject | 2
Not completed — Maintenance Therapy Screen Fail | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat))
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 61 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Toxicity of Vorinostat Bortezomib Maintenance Therapy After Autologous Transplant
Description: Number of patients on maintenance therapy post-transplant who experienced grade 3 or higher toxicity per NCI-Common Terminology Criteria for Adverse Events, version 3. The first three months of bortezomib and vorinostat therapy will be used as the time period to evaluate toxicity for stopping rules of the study. Toxicity that meets stopping rules will be determined based on the number of patients that are withdrawn from study for significant toxicity (grade IV, non-hematological, non-metabolic, non-peripheral neuropathy).
Time Frame: 3 months after start of maintenance therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat))
Number analyzed (Participants) | 19
Participants | 19

2. Secondary Outcome: Median Time to Disease Progression
Description: median days from transplant to relapse/progression
Time Frame: time post ASCT to progression
Population: median time to progression /relapse
Measure: Median (Full Range); unit: years
Arm/Group | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat))
Number analyzed (Participants) | 19
years | 1.05 [0.41 to 8.05]

3. Secondary Outcome: Ability to Complete Planned 12 Cycles of Maintenance Therapy
Description: Number of patients who completed all 12 cycles of maintenance therapy.
Time Frame: Approximately 12 months following start of maintenance therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat))
Number analyzed (Participants) | 19
Participants
  Completed 12 Cycles of Maintenance Therapy | 7
  Unable to complete therapy due to relapse | 3
  Withdrawl at patient request | 2
  Unable to complete due to toxicities | 5
  PI decision due to increasing creatinine levels | 1
  Patient left state | 1

4. Secondary Outcome: Overall Survival
Description: Number of patients alive who received maintenance therapy
Time Frame: 6.64 Years Post-Transplant
Measure: Number; unit: participants
Arm/Group | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat))
Number analyzed (Participants) | 19
participants
  Alive | 16
  Dead | 3

5. Secondary Outcome: Event-free Survival
Description: Number of patients alive without disease progression/relapse
Time Frame: 6.64 Years Post-Transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat))
Number analyzed (Participants) | 19
Participants
  Alive without disease porgression | 14
  alive with disease progression | 5

ADVERSE EVENTS:
Description: Adverse events will be evaluated according to criteria outlined in the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 3.0., except hematological toxicity. Grade 3 or higher reported.
Arm/Group | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat))
All-Cause Mortality (participants affected / at risk) | 7/27
Serious Adverse Events (participants affected / at risk) | 9/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat)) (N=27)
Atrial flutter/atrial fibrillation (Cardiac disorders) | 2 — Transplant toxicity.
Febrile neutropenia (Blood and lymphatic system disorders) | 2 — Transplant toxicity. One patient had both febrile neutropenia with transplant and pneumonia with maintenance therapy as two separate events.
Abdominal pain/diarrhea (Gastrointestinal disorders) | 1 — Maintenance therapy toxicity.
Pneumonia (Infections and infestations) | 2 — Maintenance therapy toxicity. One patient had both febrile neutropenia with transplant and pneumonia with maintenance therapy as two separate events.
Nausea, vomiting, and diarrhea requiring hospitalization (Gastrointestinal disorders) | 2 — Transplant toxicity.
Colitis (Gastrointestinal disorders) | 1 — Transplant toxicity.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Treatment (Chemotherapy, ASCT, Bortezomib, Vorinostat)) (N=27)
Anemia (Blood and lymphatic system disorders) | 3 — Autologous transplant adverse event. No patients died due to transplant therapy.
Auto GVHD (General disorders) | 2 — Autologous transplant adverse event. No patients died due to transplant therapy.
Colitis (Gastrointestinal disorders) | 2 — Autologous transplant adverse event. No patients died due to transplant therapy.
Dehydration (Metabolism and nutrition disorders) | 3 — Autologous transplant adverse event. No patients died due to transplant therapy.
Diarrhea (Gastrointestinal disorders) | 6 — Autologous transplant adverse event. No patients died due to transplant therapy.
Febrile neutropenia (Blood and lymphatic system disorders) | 21 — Autologous transplant adverse event. No patients died due to transplant therapy.
Heartburn (Gastrointestinal disorders) | 2 — Autologous transplant adverse event. No patients died due to transplant therapy.
Nausea/Vomitting (Gastrointestinal disorders) | 7 — Autologous transplant adverse event. No patients died due to transplant therapy.
Nausea (Gastrointestinal disorders) | 6 — Autologous transplant adverse event. No patients died due to transplant therapy.
Mucositis (Gastrointestinal disorders) | 16 — Autologous transplant adverse event. No patients died due to transplant therapy.
Neutropenia (Investigations) | 27 — Autologous transplant adverse event. No patients died due to transplant therapy.
Rash (Skin and subcutaneous tissue disorders) | 2 — Autologous transplant adverse event. No patients died due to transplant therapy.
Thrombocytopenia (Investigations) | 27 — Autologous transplant adverse event. No patients died due to transplant therapy.
Volume overload (General disorders) | 2 — Autologous transplant adverse event. No patients died due to transplant therapy.
Dizziness (Nervous system disorders) | 1/19 — Maintenance therapy post-transplant adverse event. No patients died due to maintenance therapy.
Hyponatremia (Metabolism and nutrition disorders) | 1/19 — Maintenance therapy post-transplant adverse event. No patients died due to maintenance therapy.
Methemoglobinemia (Blood and lymphatic system disorders) | 1/19 — Maintenance therapy post-transplant adverse event. No patients died due to maintenance therapy.
Neutropenia (Investigations) | 13/19 — Maintenance therapy post-transplant adverse event. No patients died due to maintenance therapy.
Peripheral neuropathy (Nervous system disorders) | 2/19 — Maintenance therapy post-transplant adverse event. No patients died due to maintenance therapy.
Thrombocytopenia (Investigations) | 2/19 — Maintenance therapy post-transplant adverse event. No patients died due to maintenance therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No